CLINICAL TRIAL: NCT07319585
Title: Managed Access Programs for EXV811, Atrasentan
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CEXV811A12004M
Record Dates: First submitted 2025-12-18; First posted 2026-01-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: IgA Nephropathy
Keywords: MAP; Managed Access Program; IgA Nephropathy; EXV811; Atrasentan
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Atrasentan

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Atrasentan — Patients receive atrasentan
  Other Names: EXV811

SUMMARY:
The purpose of this registration is to list Managed Access Programs (MAPs) related to EXV811, Atrasentan

DETAILED DESCRIPTION:
CEXV811A12004M - Available - Managed Access Program (MAP) Cohort Treatment Plan CEXV811A12004M to provide access to Atrasentan for IgA nephropathy

ELIGIBILITY:
Inclusion Criteria:

1. An independent request was received from a licensed physician.
2. The patient has a serious or life-threatening disease or condition and there is no comparable or satisfactory alternative therapy available for diagnosis, monitoring, or treatment.
3. The patient is not eligible or able to enrol in a clinical trial or continue participation in such trial.
4. There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
5. The patient must meet any other medical criteria established by the medical experts responsible for the product or by the health authority in the country of request (as applicable).
6. Provision of the product will not interfere with the initiation, conduct, or completion of a Novartis clinical trial or overall development program.
7. Managed Access provision is allowed per local laws/regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult